CLINICAL TRIAL: NCT05242770
Title: Feasibility of Pelvic Physical Therapy for Sexual Dysfunction in Gynecologic Oncology Survivors
Brief Title: Pelvic Physical Therapy for Sexual Dysfunction in Gynecologic Oncology Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00079802; WFBCCC 01421 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2022-01-26; First posted 2022-02-16 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2023-12

CONDITIONS: Gynecologic Cancer; Sexual Dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Placebo Comparator): Educational pamphlet with resources for sexual dysfunction
  Interventions: Other: Control Arm
- Physical Therapy Arm (Experimental): Physical therapy for sexual dysfunction.
  Interventions: Other: Physical Therapy Arm; Other: European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30); Other: Female Sexual Function Index (FSFI); Other: Exit Interview

INTERVENTIONS:
Other: Control Arm — Participants randomized to this arm will only receive educational pamphlets with resources for sexual dysfunction and will not participate in physical therapy. Participants will be contacted at 3 months and 6 months to fill out two questionnaires about sexual function and quality of life. After 6months, if participants desire a referral to physical therapy, investigators will provide a referral.
  Arms: Control Arm
Other: Physical Therapy Arm — Participants will receive a referral to begin a pelvic physical therapy regimen. Participants will complete the sexual function and quality of life questionnaires after completion of the physical therapy regimen and again 3 months after. There will be a brief exit interview.
  Arms: Physical Therapy Arm
Other: European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30) — Questionnaire designed to measure cancer patients' physical, psychological and social functions
  Arms: Physical Therapy Arm
Other: Female Sexual Function Index (FSFI) — 19-item self-report inventory designed to assess female sexual function.
  Arms: Physical Therapy Arm
Other: Exit Interview — 11-item questionnaire for participants to give feedback to investigators about teir experience with the intervention.
  Arms: Physical Therapy Arm

SUMMARY:
The purpose of this research study is to investigate the use of pelvic physical therapy for gynecologic cancer survivors who report sexual dysfunction. Physical therapy experts believe that a full 10-week regimen is necessary for true improvement of symptoms. Investigators aim to see if this tense regimen is feasible for survivors. Investigators also aim to see if patients have an improvement in their sexual function and quality of life.

DETAILED DESCRIPTION:
Primary Objective(s): To determine the feasibility of an intensive pelvic physical therapy intervention with gynecologic cancer survivors reporting sexual dysfunction. Feasibility will be determined by accrual, retention, and adherence.

Secondary Objective(s):

* To demonstrate preliminary efficacy of the pelvic physical therapy intervention on sexual function in gynecologic cancer survivors. Sexual function will be measured three times: at time of randomization (T0), after completion of the 10-week pelvic physical therapy regimen - 3 months after randomization (T1), and 3 months after T1 (T2).
* To demonstrate preliminary efficacy of the pelvic physical therapy intervention on health-related quality of life in gynecologic cancer survivors. Quality of life will be measured at three times (T0) at time of randomization, (T1) after completion of the 10-week pelvic physical therapy regimen - 3 months after randomization, and (T2) 3 months after T1

ELIGIBILITY:
Inclusion Criteria:

* History of cervical, ovarian/fallopian tube/primary peritoneal, uterine, or vulvar/vaginal cancer, regardless of stage or amount of prior therapy. Patients must have completed radiation therapy 12 weeks prior enrollment. Patients must be at least 12 weeks remote from surgery. There is no minimum time after completion of chemotherapy for enrollment. There is no upper limit of time from treatment.
* History of treatment for gynecological cancer - surgery, radiation, chemotherapy, or combination of therapies.
* Screen positive for sexual dysfunction based on answers to the Brief Sexual Symptom Checklist for Women. A patient screens positive if they answer "no" to the first question (Are you satisfied with your sexual function?) and if they select any answer other than "a" in the third question (Mark which of the following problems you are having). The other questions do not impact whether a patient screens positive or negative. They do not have an impact on study eligibility.
* English-speaking. Due to the developmental nature of this study, assessing feasibility with a small number of patients, we do not have all response tools and questionnaires translated into multiple languages. In a future larger study, it will be important to translate all documents into multiple languages in order to include non-English speakers.
* Age ≥18 years.

Exclusion Criteria:

* Active pelvic infection.
* Presence of vaginal fistula.
* Deemed not suitable for pelvic physical therapy based on physician assessment. If there is suspicion for infection, disease recurrence, or other concerning medical findings that necessitate further evaluation and work up at that time.
* Evidence of active cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-11-26 (Actual); Study Completion 2022-11-26 (Actual)

PRIMARY OUTCOMES:
Accrual to Study Intervention | At baseline
  Accrual is the number of participants that screen positive for sexual dysfunction, are eligible for entry into the study and consent to participate in the study.
Number of Participants Retained to Study Intervention | 3 months after completion of physical therapy.
  Retention is participants' attendance of pelvic physical therapy visits.
Adherence to Study Intervention | 3 months after completion of physical therapy.
  Adherence is the number of enrolled participants completing the interevention.

SECONDARY OUTCOMES:
Female Sexual Function Index (FSFI) Questionnaire | At time of randomization, 3 months after randomization and 3 months after completion of physical therapy regimen
  The questionnaire is comprised of six domains: desire [two items], arousal [four items], lubrication [four items], orgasm, satisfaction, pain [three items each]. Score range is 1 to 5. The FSFI total score is the sum of the 6 domain/subscale scores and has a maximum score of 36. Higher scores indicate better functioning. At each time point, 2-sample t-tests or Wilcoxon rank sum tests will be used to compare sexual function between groups. If feasible, mixed effects models with random intercept will be used to compare sexual function between groups over time. Intervention groups, visits, and intervention groups by visits will be included in the model. Contrasts will be used to compare sexual function between groups at each time point.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire | At time of randomization, 3 months after randomization and 3 months after completion of physical therapy regimen
  The EORTC QLQ-C30 questionnaire will be completed three times during study intervention and is patient reported to assess sexual function and health-related quality of life. Score range is 0 to 100. A high score for a functional scale represents a high/ healthy level of functioning; a high score for the global health status /quality of life represents a high quality of life; a high score for a symptom scale/item represents a high level of symptomatology / problems. At each time point, 2-sample t-tests or Wilcoxon rank sum tests will be used to compare sexual function between groups. If feasible, mixed effects models with random intercept will be used to compare sexual function between groups over time. Intervention groups, visits, and intervention groups by visits will be included in the model. Contrasts will be used to compare sexual function between groups at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Danhauer, PhD, Principal Investigator — Wake Forest Baptist Comprehensive Cancer Center; Anya Menzies, PhD, Principal Investigator — Wake Forest Baptist Comprehensive Cancer Center
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/70/NCT05242770/ICF_000.pdf